CLINICAL TRIAL: NCT06266000
Title: A Study to Compare 2 Extracts of Saw Palmetto Versus Placebo on Lower Urinary Tract Symptoms (LUTS) and Urinary Frequency
Brief Title: Comparison of 2 Extracts of Saw Palmetto Versus Placebo on Lower Urinary Tract Symptoms (LUTS) and Urinary Frequency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROPAL
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-07

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — saw palmetto extract; Palm Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Saw palmetto extract (Experimental): Saw palmetto extract taken as 2 capsules per day
  Interventions: Drug: Saw palmetto extract 320mg per day
- Comparator saw palmetto extract (Active Comparator): Commercial saw palmetto extract taken as 2 capsules per day
  Interventions: Drug: Commercial Saw palmetto extract 320mg per day
- Placebo (Placebo Comparator): Palm oil taken as 2 capsules per day
  Interventions: Drug: Palm Oil capsule

INTERVENTIONS:
Drug: Saw palmetto extract 320mg per day — Saw palmetto extract 160mg per capsule
  Arms: Saw palmetto extract
Drug: Commercial Saw palmetto extract 320mg per day — Saw palmetto extract 160mg per capsule
  Arms: Comparator saw palmetto extract
Drug: Palm Oil capsule — Palm oil capsule
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel group study to compare 2 extracts of saw palmetto versus placebo on lower urinary tract symptoms and urinary frequency in 120 generally healthy participants, 45 - 80 years.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 45-80
* Mild to moderate in the IPSS
* Generally healthy
* Able to provide informed consent
* Agree not to participate in another clinical trial while enrolled in this trial
* Agree not the change their diet or exercise while enrolled in this trial

Exclusion Criteria:

* Serious illness e.g., mood disorders such as depression, anxiety or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions (A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments)
* Unstable illness e.g., diabetes and thyroid gland dysfunction (An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity)
* Have used a drug/natural therapy for LUTS or other urological symptoms within the last 30 days?
* Have had a urinary infection in the last 30 days or have, chronic urinary tract infections, or diagnosed chronic prostatitis
* Have had urogenital surgery within the last 6 months.
* Have had a bladder biopsy and/or cystoscopy and biopsy within the past 30 days.
* Have been diagnosed with chronic persistent local pathology (e.g. interstitial cystitis, bladder stones)
* Receiving/ prescribed Coumadin (Warfarin) or other anticoagulation therapy
* Diagnosed genital anatomical deformities, uncontrolled diabetes mellitus, and history of spinal cord injury, uncontrolled psychiatric disorder, and/or abnormal secondary sexual characteristics.
* Diagnosed cancer including prostatic cancer; if suspected by the investigator, refer for medical assessment
* Active smokers and/or nicotine or drug abuse
* Chronic alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in investigational, comparator or placebo formula
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participated in any other clinical trial during the past 1 month

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Daily Urinary Frequency Log | Baseline for 7 days, Days 21-27, Day 49-55, Day 77-83
  Change from baseline to the end of the study period in Daily Urinary Frequency Diary
International Prostate Symptom Score (IPSS) | Baseline, Day 28, Day 56, Day 84
  Change from baseline to the end of the study period in the International Prostate Symptom Score (IPSS).The total score can range from 0 to 35 i.e. asymptomatic to very symptomatic.

SECONDARY OUTCOMES:
Brief Sexual Function Inventory (BSFI) | Baseline, Day 28, Day 56, Day 84
  Change from baseline to the end of the study period in Brief Sexual Function Inventory (BSFI). The total score can range from 0 to 44 with higher scores indicating better outcomes.
International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms Module (ICIQ-MLUTS) | Baseline, Day 84
  Change from baseline to the end of the study period in International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms (ICIQ-MLUTS). The total score can range from 1 to 84 with higher scores indicating worse outcomes.
Electrolytes (E/LFT) blood test | Baseline, Day 84
  Change from baseline to the end of the study period in electrolytes measured via E/LFT blood test.
Liver Function (E/LFT) blood test | Baseline, Day 84
  Change from baseline to the end of the study period in liver function measured via E/LFT blood test.
Inflammatory marker - JM27 | Baseline, Day 84
  Change from baseline to the end of the study period in Inflammatory marker - JM27 assessed via blood test
Blood pressure | Baseline, Day 84
  Change from baseline to the end of the study period in blood pressure
Pulse rate | Baseline, Day 84
  Change from baseline to the end of the study period in pulse rate
Adverse event frequency | During enrolment period
  Change in safety as assessed by adverse events frequency
Adverse event severity | During enrolment period
  Change in safety as assessed by adverse events severity
Discontinuation due to adverse events | During enrolment period
  Number of participants who discontinue study due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No